CLINICAL TRIAL: NCT05331664
Title: Dropless Pars Plana Vitrectomy Study
Acronym: DVS
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Nimesh Patel, Principal Investigator, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022P000046
Record Dates: First submitted 2022-04-09; First posted 2022-04-15 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Rhegmatogenous Retinal Detachment
Keywords: Vitrectomy; Dropless; Sub-tenon steroids; Postoperative; Inflammation; Randomized clinical trial; Non-inferiority trial
MeSH Terms: conditions — Inflammation | interventions — Triamcinolone Acetonide; Triamcinolone; Moxifloxacin; Polymyxins; 1(beta)-D-arabinofuranosylcytosine-5'-diphosphate prednisolone; prednisolone acetate; Atropine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group 1 (Active Comparator): * Subconjunctival antibiotic (cefazolin 50 mg/0.5 mL, moxifloxacin 0.5 mg/0.1 mL, or vancomycin 1 mg/0.1 mL) and subconjunctival dexamethasone (4 mg/mL) at the time of surgery
  * Topical atropine 1% and antibiotic-steroid ointment (neomycin-polymyxin B-dexamethasone) at the time of surgery
  * Topical moxifloxacin 0.5% or Polymyxin/Trimethoprim if patient is allergic to moxifloxacin; 4 times per day for 1 week after surgery.
  * Topical prednisolone 1% 1 drop 4 times per day tapered by one drop weekly for 4 weeks (4/3/2/1 taper)
  * Topical atropine 1% daily for 1 week
  Interventions: Procedure: Pars plana vitrectomy; Drug: Moxifloxacin 0.5% or Polymyxin/Trimethoprim if patient is allergic to moxifloxacin; Drug: Prednisolone 1%; Drug: Atropine 1%
- Group 2 (Active Comparator): * Subtenon triamcinolone acetonide (40 mg/1mLl) at the time of surgery
  * Subconjunctival antibiotic (cefazolin 50 mg/0.5 mL, moxifloxacin 0.5 mg/0.1 mL, or vancomycin 1 mg/0.1 mL) and subconjunctival dexamethasone (4 mg/mL) at the time of surgery
  * Topical atropine 1% and antibiotic-steroid ointment (neomycin-polymyxin B-dexamethasone) at the time of surgery
  * No postoperative eye drops
  Interventions: Procedure: Pars plana vitrectomy; Drug: Triamcinolone Acetonide 40mg/mL

INTERVENTIONS:
Procedure: Pars plana vitrectomy — Standard of care surgery
Drug: Triamcinolone Acetonide 40mg/mL — Sub-tenon injection of triamcinolone acetonide (40mg/mL) at the time of surgery
  Other Names: Kenalog-40
  Arms: Group 2
Drug: Moxifloxacin 0.5% or Polymyxin/Trimethoprim if patient is allergic to moxifloxacin — Antibiotic eye drop 4 times per day for 1 week after surgery
  Other Names: Vigamox or Polytrim
  Arms: Group 1
Drug: Prednisolone 1% — Steroid eye drop 4 times per day tapered by one drop weekly for 4 weeks (4/3/2/1 taper) after surgery
  Other Names: Pred forte
  Arms: Group 1
Drug: Atropine 1% — Eye drop daily for 1 week after surgery
  Other Names: Atropine sulfate
  Arms: Group 1

SUMMARY:
To demonstrate that intraoperative use of subtenon triamcinolone acetonide at the time of surgery without postoperative eye drops is non-inferior to the regimen of postoperative eye drops following primary pars plana vitrectomy for retinal detachment.

DETAILED DESCRIPTION:
This is a non-inferiority, single-center, randomized, controlled, open-label clinical trial. Investigators will recruit patients that present to their clinic or emergency department with newly diagnosed mac-on or mac-off rhegmatogenous retinal detachment. Patients will be randomized to one of the following groups:

* Group 1: A total of 84 study subjects (84 eyes) will receive topical antibiotic qid for one week after surgery, topical prednisolone 1% qid tapered by one drop weekly for four weeks (4/3/2/1 taper), and topical atropine 1% daily for one week.
* Group 2: A total of 84 study subjects (84 eyes) will receive sub-tenon injection of triamcinolone acetonide (40 mg/mL) at the time of surgery, with no post-operative eye drops.

Both groups will receive subconjunctival injection of antibiotic (cefazolin 50 mg/0.5 ml, moxifloxacin 0.5 mg/0.1 ml, or vancomycin 1 mg/0.1 ml) and subconjunctival injection of dexamethasone (4 mg/ml) at the time of surgery, as well as atropine 1% and antibiotic-steroid ointment (neomycin-polymyxin B-dexamethasone) at the time of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Primary rhegmatogenous retinal detachment (mac-on or mac-off) requiring pars plana vitrectomy (23, 25 and 27-gauge)

Exclusion Criteria:

* Need for concomitant lensectomy or cataract surgery
* Pars plana vitrectomy taking place more than seven days after the initial diagnosis
* History of any prior vitreoretinal surgery (excluding laser surgery) in surgical eye
* History of previous retinal detachment in surgical eye
* History of ocular incisional surgery within six months of surgery (excluding laser surgery) in surgical eye
* History of ocular laser surgery within 1 month in surgical eye
* History of intravitreal injection within 1 month in surgical eye
* Diagnosis of glaucoma or intraocular pressure more than 21 mmHg in either eye
* Active or chronic or recurrent uncontrolled ocular or systemic disease
* Active or history of chronic or recurrent inflammatory eye disease
* Previous history of steroid response
* Current treatment with oral, topical, or intravitreal corticosteroids
* Presence of proliferative vitreoretinopathy at the time of diagnosis
* Presence of giant retinal tear at the time of diagnosis
* Diagnosis of proliferative diabetic retinopathy
* Anterior chamber inflammation on presentation in either eye
* Signs of ocular infection at presentation in either eye
* Acute external ocular infections
* Known or suspected sensitivity or allergy to any of the medications used in the operation or postoperatively
* Inability to use or apply topical eye drops
* Requirement for silicone oil as a tamponade agent
* Individuals with impaired decision-making capacity
* Non-English-speaking subjects

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Estimated)
Dates: Start 2022-07-25 (Actual); Primary Completion 2026-07-25 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Mean anterior chamber cell | Day 7 after surgical procedure
  Mean anterior chamber cell based on SUN (Standardization of Uveitis Nomenclature) criteria as measured by Slit Lamp Biomicroscopy

SECONDARY OUTCOMES:
Mean anterior chamber cell | Day 1, 30 and 90 after surgical procedure
  Mean anterior chamber cell based on Standardization of Uveitis Nomenclature (SUN) criteria as measured by Slit Lamp Biomicroscopy
Need for rescue medication (corticosteroid) | Day 1, 7, 30 and 90 after surgical procedure
  Need for additional medication (corticosteroid) to control post-operative inflammation
Intraocular pressure less than 5 or more 30 mmHg | Day 1, 7, 30 and 90 after surgical procedure
  Intraocular pressure measured by applanation tonometer or tono-pen
Need for medications to reduce intraocular pressure | Day 1, 7, 30 and 90 after surgical procedure
  Need for additional medication to reduce intraocular pressure
Visual acuity | Day 1, 7, 30 and 90 after surgical procedure
  Best-corrected visual acuity measured using Snellen chart
Degree of pain | Day 1, 7, 30 and 90 after surgical procedure
  Degree of pain on a pain scale of 1-10 (0: pain free, 10: unspeakable pain)
Self-reported adherence to positioning | Day 1 and 7 after surgical procedure
  Assessment of self-reported adherence to positioning: "Over the past day or week, what percentage of time or number of hours per day do you think you adhered with the recommended positioning?"
Self-reported adherence to eye drops | Day 1, 7 and 30 after surgical procedure
  Assessment of self-reported adherence to eye drops in the control group: "Over the past week or month, what percentage of your drops do you think you took correctly?"
Progression of cataract | Day 30 and 90 after surgical procedure
  Evaluation of progression of cataract by Slit Lamp Biomicroscopy
Adverse events | Day 1, 7, 30 and 90 after surgical procedure
  Adverse Events including: Endophthalmitis, Re-detachment requiring surgery, Intraocular pressure requiring medication, Need for additional procedures, Any other adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Nimesh A. Patel, MD, Principal Investigator — Massachusetts Eye and Ear
Locations (1):
- Massachusetts Eye and Ear, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paccola L, Jorge R, Barbosa JC, Costa RA, Scott IU. Anti-inflammatory efficacy of a single posterior subtenon injection of triamcinolone acetonide versus prednisolone acetate 1% eyedrops after pars plana vitrectomy. Acta Ophthalmol Scand. 2007 Sep;85(6):603-8. doi: 10.1111/j.1600-0420.2007.00923.x. Epub 2007 Apr 24. PMID 17459031
- [Background] Brown GT, Karth PA, Hunter AA. Novel Postoperative Dropless Protocol for Micro-Incision Vitrectomy Surgery. Ophthalmic Surg Lasers Imaging Retina. 2021 Nov;52(11):587-591. doi: 10.3928/23258160-20211014-01. Epub 2021 Nov 1. PMID 34766851
- [Background] Bonfiglio V, Reibaldi M, Macchi I, Fallico M, Pizzo C, Patane C, Russo A, Longo A, Pizzo A, Cillino G, Cillino S, Vadala M, Rinaldi M, Rejdak R, Nowomiejska K, Toro MD, Avitabile T, Ortisi E. Preoperative, Intraoperative and Postoperative Corticosteroid Use as an Adjunctive Treatment for Rhegmatogenous Retinal Detachment. J Clin Med. 2020 May 21;9(5):1556. doi: 10.3390/jcm9051556. PMID 32455658
- [Background] Assil KK, Greenwood MD, Gibson A, Vantipalli S, Metzinger JL, Goldstein MH. Dropless cataract surgery: modernizing perioperative medical therapy to improve outcomes and patient satisfaction. Curr Opin Ophthalmol. 2021 Jan;32 Suppl 1:S1-S12. doi: 10.1097/ICU.0000000000000708. PMID 33273209
- See also: A retrospective consecutive case series showing that single subconjunctival triamcinolone acetonide injection at the end of surgery may represent a reasonable alternative to requiring patients to use a steroid drop taper following vitreoretinal surgery. — https://www.semanticscholar.org/paper/Elimination-of-Steroid-Drops-After-Vitreoretinal-Atchison-Gilca/e5b33498c8b088eb6538feb612e20b6d220705f1